CLINICAL TRIAL: NCT01552707
Title: "Ex Vivo" Expanded Autologous Bone Marrow Mesenchymal Stem Cells Fixed in Allogenic Human Bone Tissue for Spinal Fusion in Spine Degenerative Disease
Brief Title: Safety Study of Mesenchymal Stem Cells and Spinal Fusion
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Banc de Sang i Teixits (Other)
Collaborators: TFS Trial Form Support (Industry); Ministerio de Sanidad, Servicios Sociales e Igualdad (Other Government); Ministerio de Ciencia e Innovación, Spain (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XCEL-MT-10-02
Record Dates: First submitted 2012-03-08; First posted 2012-03-13 (Estimated); Last update posted 2020-01-21 (Actual); Status verified 2020-01

CONDITIONS: Lumbar Spondylolisthesis Involving L4-L5, and/or; Degenerative Discopathy Involving L4-L5
Keywords: Spondylolisthesis; Degenerative discopathy; Mesenchymal Stem Cells; Bone marrow; Tissue engineering; Spinal fusion
MeSH Terms: conditions — Spondylolisthesis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- XCEL-MT-OSTEO-ALPHA (Experimental): "ex-vivo" expanded autologous mesenchymal stem cells fixed in allogenic bone tissue for spinal fusion
  Interventions: Biological: XCEL-MT-OSTEO-ALPHA
- Standard treatment (Sham Comparator): Instrumented spinal fusion together with patient's bone iliac crest.
  Interventions: Procedure: Standard treatment

INTERVENTIONS:
Biological: XCEL-MT-OSTEO-ALPHA — Isolation and "ex-vivo" expansion of mesenchymal stem cells (MSC) obtained from each patient's bone marrow under GMP conditions at Xcelia, División de Terapias Avanzadas delBanc de Sang i Teixits. After expansion, MSCs are fixed in allogenic bone tissue and implanted in instrumented spinal fusion.
  Arms: XCEL-MT-OSTEO-ALPHA
Procedure: Standard treatment — Instrumented spinal fusion together with patient's bone iliac crest
  Arms: Standard treatment

SUMMARY:
The present prospective, randomized study, compares the spinal fusion obtained after instrumentation and the use of a biologic product (patient's mesenchymal cells obtained from his/her own bone marrow which will be fixed in human bone tissue form a donor), with the current procedure that consists in instrumented spinal fusion and the use of each patient's bone obtained from his/her iliac crest.

The working hypothesis proposes that the tissue engineering is a valid and useful technique to achieve bone regeneration, avoiding the need for obtaining patient's iliac crest and its associated morbidity.

DETAILED DESCRIPTION:
Prospective, open-label, randomized, parallel, single-dose phase I-II clinical trial in which 62 patients affected with L4-L5 degenerative spondylolisthesis grade I-II according to Meyerding and/or with L4-L5 degenerative discopathy needing spinal fusion will enter the trial with the primary objective of assessing the feasibility and safety of "ex-vivo" expanded autologous mesenchymal stem cells fixed in allogenic bone tissue in spinal fusion. Secondary objectives are to assess the efficacy of the implantation by imaging (computerized helicoidal tomography and X-ray) and clinical questionnaires (pain by visual analogue scale, quality of life by SF-36 and Oswestry Disability Index).

Patients will be randomized to one of the two treatment arms (instrumented spinal fusion and the tissue engineering product composed by "ex-vivo" expanded autologous mesenchymal stem cells fixed in allogenic bone tissue in spinal fusion or the standard treatment of instrumented spinal fusion and patient's bone iliac crest). Thereafter, patients will be followed for 12 months.

Imaging assessment will be done by an independent blinded radiologist.

ELIGIBILITY:
Inclusion Criteria:

* L4-L5 degenerative spondylolisthesis grade I-II Meyerding isolated or associated to more than one level, and/or L4-L5 degenerative discopathy isolated or associated to more than one level.
* 18 to 85 years of age (male and female)
* Informed Consent Form signed
* The patient is able to understand the nature of the study

Exclusion Criteria:

* Previous spine surgery
* L4 isthmic spondylolisthesis
* Smoker (more than 10 cigarettes a day)
* Systemic or local infection
* Patients treated with steroids (oral or systemic) within 3 months of entering the study, or treated with biphosphonates for more than 10 years
* Positive serology for HIV-1 or HIV-2, Hepatitis B (HBsAg), Hepatitis C (Anti-HCV-Ab) or Syphilis.
* Pregnant woman or intended to become pregnant, or breath feeding
* Neoplasia within the previous 5 years, or without remission
* Immunosuppressive states (except diabetes mellitus. Treatment with therapies is allowed)
* Significant abnormal laboratory tests that contraindicates the surgery.
* Participation in another clinical trial or treated with an investigational medicinal product the previous 3 months
* Other pathologic conditions or circumstances that difficult participation in the study according to medical criteria
* The patient does not accept to be followed-up for a period that could exceed the clinical trial length
* The patient is legally dependent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2012-07-19 (Actual); Primary Completion 2018-05-03 (Actual); Study Completion 2019-10-21 (Actual)

PRIMARY OUTCOMES:
safety of XCEL-MT-OSTEO-ALPHA (tissue engineering product composed by "ex-vivo" expanded autologous mesenchymal stem cells fixed in allogenic bone tissue in spinal fusion) | 12 months
  Safety will be assessed by collecting adverse events throughout the experimental phase, which includes a follow-up of 12 months
Feasibility of XCEL-MT-OSTEO-ALPHA (composed by "ex-vivo" expanded autologous mesenchymal stem cells fixed in allogenic bone tissue in spinal fusion) | 12 months
  Feasibility will be measured by assessing the percentage of patients to which bone marrow puncture is made are thereafter treated and by checking the cascade of procedures to confirm the global process is viable.

SECONDARY OUTCOMES:
Efficacy spinal fusion by imaging procedures (X-Ray). | 3, 6 and 12 months
  Spinal fusion will be assessed by spinal X-Ray
Efficacy spinal fusion by imaging procedures (computerized helicoidal tomography) | 6 and 12 months
  Spinal fusion will be assessed by the presence of solid bonny bridges using computerized helicoidal tomography.
Clinical outcomes (VAS) | 7 days and at 3, 6 and 12 months
  Pain measurement by visual analogue scale (VAS)
Clinical outcomes (SF-36) | 3, 6 and 12 months
  This clinical outcome will measure the quality of life by the self-reported quality of life questionnaire SF-36
Clinical outcome (Oswestry Disability Index) | 3, 6 and 12 months
  To assess the extent by which a person's functional level is restricted by disability by the Oswestry Disability Index

CONTACTS AND LOCATIONS:
Overall Officials: Joan Bagó, MD, PhD, Principal Investigator — Hospital Vall d'Hebron
Locations (5):
- Spain (5):
  - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Parc de Salut Mar, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Institut Universitari Dexeus (ICATME), Barcelona
  - Hospital Vall d'Hebron, Barcelona

REFERENCES:
- [Derived] Vives J, Oliver-Vila I, Pla A. Quality compliance in the shift from cell transplantation to cell therapy in non-pharma environments. Cytotherapy. 2015 Aug;17(8):1009-14. doi: 10.1016/j.jcyt.2015.02.002. Epub 2015 Mar 10. PMID 25769789
- See also: Banc de Sang i Teixits. Xcelia, División de Terapias Avanzadas. — http://www.bancsang.net
- See also: Institut Català de Traumatologia i Medicina de l'Esport (Institut Universitari Dexeus) — http://www.icatme.com
- See also: Hospital Universitari Vall d'Hebron, Barcelona — http://www.vhebron.net
- See also: Hospital Universitari Germans Trias i Pujol, Badalona — http://www.gencat.cat/ics/germanstrias/
- See also: Hospital Parc de Salut Mar, Barcelona — http://www.parcdesalutmar.cat
- See also: Hospital de la Santa Creu i Sant Pau, Barcelona — http://www.santpau.es/